CLINICAL TRIAL: NCT06367309
Title: ExtrAperitoneaL Plasty vs Intraperitoneal oNlay mEsh in Ventral Hernia Repair - the Randomized Controlled ALPINE Trial
Brief Title: ExtrAperitoneaL Plasty vs Intraperitoneal oNlay mEsh in Ventral Hernia Repair
Acronym: ALPINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: St. Clara Hospital, Basel, Switzerland (Unknown); Innklinikum Altötting, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023 - 02357
Record Dates: First submitted 2024-03-27; First posted 2024-04-16 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Ventral Hernia; Abdominal Wall Defect
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The trial participants and the assessors (trained investigators not involved in the operative procedures) of the primary outcome are blinded regarding the performed procedure during the first seven days after the procedure to reduce bias. The blinding is guaranteed by not sharing the detailed operation report with anyone involved in the aftercare of the patient or in the assessment of study outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTEP (Extended totally extraperitoneal repair) (Experimental): The anterior rectus sheath is incised and the retromuscular space is entered through the rectus muscle fibres. The capnopreperitoneum is established and blunt dissection of the retromuscular space is performed. Two additional laparoscopic ports are established 8-10cm lateral to the linea alba caudally to the initial port. The medial border of the rectus sheath is incised and the preperitoneal space below the linea alba is dissected. The hernia orifice is also dissected from peritoneum and preperitoneal fatty tissue. The medial border of the right retromuscular space is then incised and blunt dissection is performed. The hernia orifice is closed with barbed suture and a synthetic mesh is placed on the posterior sheath of the dissected space (intended Mesh-defect ratio 16). The mesh is fixed non-traumatically using glubran glue or no fixation at all.
  Interventions: Procedure: Extended totally extraperitoneal repair
- IPOM (intraperitoneal onlay mesh) (Active Comparator): Capnoperitoneum is established through left sided subcostal Veress-Needle punction. Three laparoscopic ports are placed 8-10cm lateral to the linea alba usually on the patient's left side. The peritoneum is incised and detached from the umbilical and supraumbilical linea alba. The peritoneum including the hernia sac and preperitoneal fat is resected. The hernia orifice is then closed using a barbed suture. A coated mesh is than placed to the ventral abdominal wall covering the closed hernia orifices (intended mesh-defect-ratio: 16). The mesh is fixed with two transfacial absorbable sutures and several absorbable tackers placed in double crown technique around the hernia orifice. The capnoperitoneum is released, the trocars removed and the fascia closed with an absorbable suture. The skin is sutured with absorbable sutures.
  Interventions: Procedure: Intraperitoneal onlay mesh

INTERVENTIONS:
Procedure: Extended totally extraperitoneal repair — The anterior rectus sheath is incised and the retromuscular space is entered through the rectus muscle fibres. The capnopreperitoneum is established and blunt dissection of the retromuscular space is performed. Two additional laparoscopic ports are established 8-10cm lateral to the linea alba caudally to the initial port. The medial border of the rectus sheath is incised and the preperitoneal space below the linea alba is dissected. The hernia orifice is also dissected from peritoneum and preperitoneal fatty tissue. The medial border of the right retromuscular space is then incised and blunt dissection is performed. The hernia orifice is closed with barbed suture and a synthetic mesh is placed on the posterior sheath of the dissected space (intended Mesh-defect ratio 16). The mesh is fixed non-traumatically using glubran glue or no fixation at all.
  Arms: eTEP (Extended totally extraperitoneal repair)
Procedure: Intraperitoneal onlay mesh — Capnoperitoneum is established through left sided subcostal Veress-Needle punction. Three laparoscopic ports are placed 8-10cm lateral to the linea alba usually on the patient's left side. The peritoneum is incised and detached from the umbilical and supraumbilical linea alba. The peritoneum including the hernia sac and preperitoneal fat is resected. The hernia orifice is then closed using a barbed suture. A coated mesh is than placed to the ventral abdominal wall covering the closed hernia orifices (intended mesh-defect-ratio: 16). The mesh is fixed with two transfacial absorbable sutures and several absorbable tackers placed in double crown technique around the hernia orifice. The capnoperitoneum is released, the trocars removed and the fascia closed with an absorbable suture. The skin is sutured with absorbable sutures.
  Arms: IPOM (intraperitoneal onlay mesh)

SUMMARY:
This study investigates on the effect of two different operative techniques to treat abdominal wall hernias.

The goal of this clinical trial is to learn if the eTEP (Extended totally extraperitoneal repair) technique leads to a better outcome than the IPOM (Intraperitoneal onlay mesh) technique.

The main questions it aims to answer are:

* pain after the operation
* rate of complications
* rate of recurrence and reoperations
* quality of life.

Participants will:

Either be operated using the eTEP or the IPOM technique. Be followed up either in person or via email / phone call at day 1, day 7, day 14, 6 weeks, 6 months, 1, 3 and 5 years after the surgery to asses the above-stated main and some more outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years
* Informed consent obtained
* Primary or incisional ventral hernia
* Epigastric, umbilical or infraumbilical ventral hernias with transversal diameter >1cm and </= 4cm, +/- rectus diastasis which doesn't demand specific treatment
* If multiple hernias: cumulative transversal diameter </= 4cm
* Considered eligible for minimally-invasive approach

Exclusion Criteria:

* Subxyphoidal or suprapubic hernias
* precedent hernia treatment with mesh placement in the retromuscular space
* liver disease defined by the presence of ascites
* end-stage renal disease requiring dialysis
* need of an emergency surgery
* pregnancy
* need of rectus diastasis treatment intraoperatively

Criteria for participating surgeons

- Each participating surgeon has performed 20 or more laparoscopic IPOM procedures and 20 or more eTEP procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
primary outcome: pain numeric rating scale (NRS) | 24 hours
  pain, measured on the numeric rating scale (NRS) 0 - 10 24 hours after the surgical procedure.
pain outcome using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity Short Form 3a | 24 hours
  pain, measured using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity Short Form 3a 24 hours after the surgical procedure

SECONDARY OUTCOMES:
pain mid-term | 12 months
  pain, measured on the visual analog scale (NRS) 0 - 10 and using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity Short Form 3a after 7days, 14 days, 6 weeks, 6 and 12 months (NRS 0-10)
recurrence and reoperation | 5 years
  Long-term outcome at 3 and 5 years with assessment of the number of patients with clinical and / or radiological recurrences and with assessment of the number of patients who needed reoperations for either recurrences or other reasons such as mechanical bowel obstructions
LOS | 30 days
  Length of hospital stay
Functional recovery | 5 years
  Functional recovery measured using the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire at 7 and 14 days, 6 weeks, 6 months, 1, 3 and 5 years.
  The questionnaire uses 5 questions describing the patients health & abilities on that particular day and a visual analogue scale question (0 = worst, 100 = best) on the patients health on that particular day.
Adverse events | 30 days
  Intraoperative adverse events (Bleeding, conversion rate, injury to bowel structures) Postoperative adverse events (ileus, seroma, hematoma, Surgical site infections (SSI), pulmonary embolism) according to Clavien-Dindo Classification and scored according to the Comprehensive Complication Index (CCI) up to 30 days after surgery.
Quality of life (SF 12) | 5 years
  Quality of life using the short form-12 (SF-12) questionnaire at 7 and 14 days, 6 weeks, 6 months, 1, 3 and 5 years.
  The 12-item Short Form Survey (SF-12) is a general health questionnaire that was first published in 1995 as part of the Medical Outcomes Study (MOS). The SF-12 was constructed using questions drawn from each of the 8 dimensions of the MOS 36 item Short Form Survey (SF-36).
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12).
  The score ranges from 0 - 100, with a higher score indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Süsstrunk, MD, Principal Investigator — Clarunis - Universitäres Bauchzentrum Basel; Johannes Baur, MD, Principal Investigator — Clarunis - Universitäres Bauchzentrum Basel
Locations (1):
- St. Clara Hospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared upon reasonable request. Only anonymised data shall be shared.